CLINICAL TRIAL: NCT00991991
Title: Identification of Genomic Lesions Promoting Nodal Metastasis in Malignant Melanoma
Brief Title: Study of Tumor Tissue Samples From Patients With Stage I, Stage II, or Stage III Malignant Melanoma
Status: Terminated | Type: Observational
Why Stopped: Not enough tissue for analysis
Sponsor: Case Comprehensive Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CASE1609; P30CA043703 (NIH); CASE1609 (Other: Case Comprehensive Cancer Center); CASE 1609-CC733 (Other: Cancer Center IRB)
Record Dates: First submitted 2009-10-07; First posted 2009-10-08 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Melanoma (Skin)
Keywords: stage I melanoma; stage II melanoma; stage III melanoma
MeSH Terms: conditions — Melanoma | interventions — Gene Expression Profiling; Polymerase Chain Reaction; Amplified Fragment Length Polymorphism Analysis

STUDY DESIGN:
Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — tumor tissue samples from patients with stage I, stage II, or stage III malignant melanoma
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Genetic: gene expression analysis — Laser capture microdissection is performed on the archived tissue samples to isolate melanoma cells. DNA is then purified from the samples and amplified using PCR. Matrix-assisted laser desorption/ionization (MALDI)-time of flight mass spectrometry technology is used to detect mutations of B-Raf and N-Ras. Single nucleotide polymorphism arrays are also performed.
Genetic: polymerase chain reaction — Laser capture microdissection is performed on the archived tissue samples to isolate melanoma cells. DNA is then purified from the samples and amplified using PCR. Matrix-assisted laser desorption/ionization (MALDI)-time of flight mass spectrometry technology is used to detect mutations of B-Raf and N-Ras. Single nucleotide polymorphism arrays are also performed.
Genetic: polymorphism analysis — Laser capture microdissection is performed on the archived tissue samples to isolate melanoma cells. DNA is then purified from the samples and amplified using PCR. Matrix-assisted laser desorption/ionization (MALDI)-time of flight mass spectrometry technology is used to detect mutations of B-Raf and N-Ras. Single nucleotide polymorphism arrays are also performed.
Other: matrix-assisted laser desorption/ionization time of flight mass spectrometry — Laser capture microdissection is performed on the archived tissue samples to isolate melanoma cells. DNA is then purified from the samples and amplified using PCR. Matrix-assisted laser desorption/ionization (MALDI)-time of flight mass spectrometry technology is used to detect mutations of B-Raf and N-Ras. Single nucleotide polymorphism arrays are also performed.
Other: medical chart review — Information about the patient's demographics (e.g., TNM staging, sex, age, and tissue collection dates) will be gathered by chart review or from the Multidisciplinary Melanoma Conference at University Hospitals tumor conference report in order to match cases.

SUMMARY:
RATIONALE: Studying the genes expressed in samples of tumor tissue from patients with cancer may help doctors identify biomarkers related to cancer.

PURPOSE: This research study is looking at tumor tissue samples from patients with stage I, stage II, or stage III malignant melanoma.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the genetic profile of primary melanomas with and without synchronous regional nodal involvement by examining for 1) activating mutations B-Raf and N-Ras associated with melanoma development, and 2) allelic imbalances across the genome.
* Compare the genetic profile of primary melanomas from patients with and without lymph node involvement.
* Determine the combinations of genetic lesions that correlate with nodal metastasis by adopting a statistical machine learning approach to build a lesion-based classifier for nodal metastasis.

OUTLINE: Laser capture microdissection is performed on the archived tissue samples to isolate melanoma cells. DNA is then purified from the samples and amplified using PCR. Matrix-assisted laser desorption/ionization (MALDI)-time of flight mass spectrometry technology is used to detect mutations of B-Raf and N-Ras. Single nucleotide polymorphism arrays are also performed.

Information about the patient's demographics (e.g., TNM staging, sex, age, and tissue collection dates) will be gathered by chart review or from the Multidisciplinary Melanoma Conference at University Hospitals tumor conference report in order to match cases.

ELIGIBILITY:
Inclusion Criteria:

* Node positive Group (experimental group)

  * Primary melanoma > 2 mm in depth
  * Metastasis must be > 0.1 mm and detectable by IHC or hematoxylin and eosin (H&E) to be considered node positive
  * Slides and block for primary and node must be archived in UH dermatopathology
* Node Negative Group (control group)

  * Primary melanoma > 2 mm in depth
  * A negative sentinel lymph node must be negative by IHC and H&E

    * No stage IV disease
    * No acral and mucosal histology
    * No history of prior invasive melanoma
    * Underwent primary excision and sentinel lymph node biopsy within 3 months of each other
    * Archived tissue available
  * Slides and block for primary tumor and node biopsy must be archived in University Hospitals Case Medical Center (UH) dermatopathology

Exclusion Criteria:

* Acral and mucosal histology
* Previous diagnosis of invasive melanoma
* previous chemotherapy or immunotherapy
* patients who are found to have stage IV disease during workup

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Tumor tissue samples from patients with stage I, stage II, or stage III malignant melanoma. Primary care clinic
Sampling Method: Probability Sample
Enrollment: 5 (Actual)
Dates: Start 2009-07; Primary Completion 2016-03 (Actual); Study Completion 2016-03 (Actual)

PRIMARY OUTCOMES:
Genetic profile of patients with primary melanomas with and without synchronous regional nodal involvement | at the time of presentation
Comparison of genetic profile of patients with primary melanomas with and without synchronous regional nodal involvement | at the time of presentation
Combinations of genetic lesions that correlate with nodal metastasis | at the time of presentation

CONTACTS AND LOCATIONS:
Overall Officials: Henry Koon, MD, Principal Investigator — Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center
Locations (1):
- Case Medical Center, University Hospitals Seidman Cancer Center, Case Comprehensive Cancer Center, Cleveland, Ohio, United States